CLINICAL TRIAL: NCT04592770
Title: Effect of Nature-based Exercise on Post-traumatic Growth Among People With Post-traumatic Stress: A Randomized Placebo-controlled Trial Designed to Observe Psychophysiological Alterations Before to After Intervention
Brief Title: Effect of Exercise on Post-traumatic Growth Among Health Care Providers With Post-traumatic Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Karachi (Other)
Responsible Party: Principal Investigator, Shamoon Noushad, Principal Investigator, University of Karachi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KU-DoHPESS-5
Record Dates: First submitted 2020-10-01; First posted 2020-10-19 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Post Traumatic Stress Disorder
Keywords: natural environment; walking; post traumatic growth; traumatic stress
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — 4-Acetamido-4'-isothiocyanatostilbene-2,2'-disulfonic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The experimental intervention (walk): (Experimental): In this group, the nature walk will take place in a conserved and by far the largest recreational area of Karachi city. The safari park covering an area of 148 acres (0.60 km2), It has a zoo, geared with woodland, mountain viewing, safari tracks, as well as two natural lakes. The experiment will take place in the afternoon on a 5 km marked area. The duration of the stretching exercise sessions will be of 10 minutes followed by 50 minutes' walk session five times per week (total 12 weeks). participants will be asked to walk at moderate pace.
  Interventions: Behavioral: Nature based walk therapy
- The control intervention (sit & relax): (Placebo Comparator): Subjects will undergo 12 weeks of nature therapy that includes exposure to natural landscapes. The duration of the sessions will be 60 minutes five times per week. The subjects will be asked to sit and relax in the evening, in the same recreational area which is used for the experimental group.
  Interventions: Behavioral: Sit in nature

INTERVENTIONS:
Behavioral: Nature based walk therapy — 10 minutes stretching exercises followed by walk in nature for 50 minutes
  Other Names: Experimental
  Arms: The experimental intervention (walk):
Behavioral: Sit in nature — Sit in nature for 60 minutes
  Other Names: Control
  Arms: The control intervention (sit & relax):

SUMMARY:
The purpose of designing this randomized control trial is to observe the effect of nature-based walk on post-traumatic growth and Psychophysiological alterations associated with it, in traumatic stress among health care providers of Karachi Pakistan. This study is planned to investigate the recreational exposure to the natural environment for the promotion of PTG, in the traumatic stress subjects and to determine whether PTG is associated with psychophysiological alterations, i.e. C-Reactive Protein, Brain Derived Neurotropic Factor, Interleukin-6, Cortisol, and Heart Rate Variability. Subjects who had experienced any traumatic event in the last 12 months will be recruited, and at baseline, the participant will be assessed with Trauma Symptom Checklist 40 to evaluate trauma intensity. Moreover, subjects who had developed PTG or did not have any trauma intensity will be excluded from the study. Blinded treatment will be provided to subjects meeting eligibility criteria and will be randomized into two groups sequentially as they agree to participate. The nature-based walk will be used as intervention vs the control (relax in nature). The study outcomes will be monitored in subjects of both groups at different intervals, i.e. at baseline and 3-month follow-up (post-interventional).

DETAILED DESCRIPTION:
Plan of work

* Enrollment: Those subjects who had experienced any traumatic event in the last 12 months will be enrolled.
* Assessment of eligibility: Subject meeting eligibility criteria will be included in the study.
* Baseline assessment: All the variables, i.e. Post-traumatic growth inventory (PTGI), Trauma symptom checklist-40 (TSC-40), Traumatic stress scale (TSS), C-Reactive protein (CRP), Brain-derived neurotrophic factor (BDNF), Interleukin-6 (IL-6), Cortisol and Heart rate variability (HRV) will be measured at baseline.
* Randomization: Subjects based on eligibility criteria will be randomly allocated to the experimental or control group sequentially as they agree to participate.
* Allocation: A booklet with detailed instructions will be provided to the study subjects according to the groups allocated.
* Follow-up assessment: After 3 months, all the variables measured at the baseline phase will be measured again.
* Statistical Analysis: Pre & post-analysis will be conducted in this phase.

Participants Subjects for the present study will be recruited from 5 Health care organizations based in Karachi, Pakistan. The targeted population includes subjects from diverse ethnicity and considered eligible for participation in the study if they indicated in a pre-screening form that they had experienced a traumatic event. These subjects will be invited to participate in the study through advertisements on the notice board of each center. Written informed consent will be obtained from each study subject after providing detailed information regarding the objectives of the study and its duration.

Randomization Subjects based on eligibility criteria will be randomly allocated to the experimental or control group in the 1:1 ratio. Computer-generated random numbers will be used for randomization. After taking the subject's basic information, a unique code will be provided to each included subject by the study center. The code will be mentioned in each form of each subject.

Interventions • The experimental intervention: In this group, the nature walk will take place in a conserved and by far the largest recreational area of Karachi city. The safari park covering an area of 148 acres (0.60 km2), It has a zoo, geared with woodland, mountain viewing, safari tracks, as well as two natural lakes. The experiment will take place in the afternoon on a 5 km marked area. The duration of the stretching exercise sessions will be of 10 minutes followed by 50 minutes' walk session five times per week (total 12 weeks). participants will be asked to walk at moderate pace.

• The control intervention: Subjects will undergo 12 weeks of nature therapy that includes exposure to natural landscapes. The duration of the sessions will be 60 minutes five times per week. The subjects will be asked to sit and relax in the evening, in the same recreational area which is used for the experimental group.

ELIGIBILITY:
Inclusion Criteria:

1. Both genders, aged 16-50 years
2. Must be disease free (by their reports), there must be no evidence of any metastatic disease.
3. Fluent in written and spoken the Urdu language (National Language of Pakistan).
4. Experienced any traumatic event in the last 12 months.
5. Informed written consent
6. Being able to walk five times per week. (Participants will be asked to complete the Physical Activity Readiness Questionnaire)

Exclusion Criteria:

1. Subjects who received a structured psychological intervention for at least six months during the last three years performed by a psychologist or psychiatrist will be excluded.
2. Those with a codified psychiatric disorder (according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V) who received Psychopharmacological treatment during the last three years will also be excluded from the study sample.
3. Those subjects who had developed Post Traumatic Growth. (will be evaluated from Post Traumatic Growth Inventory)
4. Those subjects who do not have any trauma intensity. (will be evaluated from Trauma Symptom Checklist 40)
5. Subjects who are at high risk for physical injury during exercise.
6. Self-reported current and regular exercise in nature

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 246 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2021-08-10 (Actual)

PRIMARY OUTCOMES:
Post-Traumatic Growth (PTG) | 3 Months
  Change in post-traumatic growth from baseline to post-intervention assessment. Post-Traumatic Growth Inventory will be used to assess this outcome. This inventory is comprising of 21 questions based on 5 factors i.e. spiritual modifications, self-conception and alterations in viewpoints, relationship changes, new motivations and interests in life and the discovery of individual resources attainable by themselves and others. Likert scale will be used for rating where 0 means no change experienced, to increasing consequently as 5 means change experienced to a greater degree.
Traumatic Stress | 3 Months
  Change in traumatic Stress from baseline to post-intervention assessment. trauma symptom checklist - 40 will be used to assess this outcome. This 40-item instrument measure assesses trauma-related problems in categories like Dissociation, Anxiety, Depression, SATI (Sexual Abuse Trauma Index), Sleep Disturbance & Sexual Problems. using a four point scale ranging from 0 means never, to 3 means often.

SECONDARY OUTCOMES:
C- Reactive Protein (CRP) | 3 Months
  Change in the CRP level will be observed among the subjects enrolled in the experimental group as compared to the control group
Brain-derived neurotrophic factor (BDNF) | 3 Months
  Change in the BDNF level will be observed among the subjects enrolled in the experimental group as compared to the control group
Interleukin-6 (IL-6) | 3 Months
  Change in the IL-6 level will be observed among the subjects enrolled in the experimental group as compared to the control group
Cortisol | 3 Months
  Change in the cortisol level will be observed among the subjects enrolled in the experimental group as compared to the control group

OTHER OUTCOMES:
Heart Rate Variability (HRV) | 3 Months
  Change in the HRV will be observed among the subjects enrolled in the experimental group as compared to the control group

CONTACTS AND LOCATIONS:
Overall Officials: Basit Ansari, Ph.D, Study Chair — University of Karachi; Sadaf Ahmed, Ph.D, Study Director — University of Karachi
Locations (1):
- Shamoon Noushad, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alper B, Erdogan B, Erdogan MO, Bozan K, Can M. Associations of Trauma Severity with Mean Platelet Volume and Levels of Systemic Inflammatory Markers (IL1beta, IL6, TNFalpha, and CRP). Mediators Inflamm. 2016;2016:9894716. doi: 10.1155/2016/9894716. Epub 2016 Apr 5. PMID 27127347
- [Background] Brown DK, Barton JL, Gladwell VF. Viewing nature scenes positively affects recovery of autonomic function following acute-mental stress. Environ Sci Technol. 2013 Jun 4;47(11):5562-9. doi: 10.1021/es305019p. Epub 2013 May 16. PMID 23590163
- [Background] Gladwell VF, Brown DK, Barton JL, Tarvainen MP, Kuoppa P, Pretty J, Suddaby JM, Sandercock GR. The effects of views of nature on autonomic control. Eur J Appl Physiol. 2012 Sep;112(9):3379-86. doi: 10.1007/s00421-012-2318-8. Epub 2012 Jan 21. PMID 22270487
- [Background] Gladwell VF, Brown DK, Wood C, Sandercock GR, Barton JL. The great outdoors: how a green exercise environment can benefit all. Extrem Physiol Med. 2013 Jan 3;2(1):3. doi: 10.1186/2046-7648-2-3. PMID 23849478
- [Background] Hartig T, Mitchell R, de Vries S, Frumkin H. Nature and health. Annu Rev Public Health. 2014;35:207-28. doi: 10.1146/annurev-publhealth-032013-182443. Epub 2014 Jan 2. PMID 24387090
- [Background] Kerai SM, Khan UR, Islam M, Asad N, Razzak J, Pasha O. Post-traumatic stress disorder and its predictors in emergency medical service personnel: a cross-sectional study from Karachi, Pakistan. BMC Emerg Med. 2017 Aug 29;17(1):26. doi: 10.1186/s12873-017-0140-7. PMID 28851280
- [Background] Kondo MC, Fluehr JM, McKeon T, Branas CC. Urban Green Space and Its Impact on Human Health. Int J Environ Res Public Health. 2018 Mar 3;15(3):445. doi: 10.3390/ijerph15030445. PMID 29510520
- [Background] Britton E, Kindermann G, Domegan C, Carlin C. Blue care: a systematic review of blue space interventions for health and wellbeing. Health Promot Int. 2020 Feb 1;35(1):50-69. doi: 10.1093/heapro/day103. PMID 30561661
- [Background] Li Q, Otsuka T, Kobayashi M, Wakayama Y, Inagaki H, Katsumata M, Hirata Y, Li Y, Hirata K, Shimizu T, Suzuki H, Kawada T, Kagawa T. Acute effects of walking in forest environments on cardiovascular and metabolic parameters. Eur J Appl Physiol. 2011 Nov;111(11):2845-53. doi: 10.1007/s00421-011-1918-z. Epub 2011 Mar 23. PMID 21431424
- [Background] Michopoulos V, Norrholm SD, Jovanovic T. Diagnostic Biomarkers for Posttraumatic Stress Disorder: Promising Horizons from Translational Neuroscience Research. Biol Psychiatry. 2015 Sep 1;78(5):344-53. doi: 10.1016/j.biopsych.2015.01.005. Epub 2015 Jan 30. PMID 25727177
- [Background] Ohly H, White MP, Wheeler BW, Bethel A, Ukoumunne OC, Nikolaou V, Garside R. Attention Restoration Theory: A systematic review of the attention restoration potential of exposure to natural environments. J Toxicol Environ Health B Crit Rev. 2016;19(7):305-343. doi: 10.1080/10937404.2016.1196155. Epub 2016 Sep 26. PMID 27668460
- [Background] Valtchanov D, Barton KR, Ellard C. Restorative effects of virtual nature settings. Cyberpsychol Behav Soc Netw. 2010 Oct;13(5):503-12. doi: 10.1089/cyber.2009.0308. Epub 2010 Feb 25. PMID 20950174
- [Background] Noushad S, Ahmed S, Ansari B, Mustafa UH, Saleem Y, Hazrat H. Physiological biomarkers of chronic stress: A systematic review. Int J Health Sci (Qassim). 2021 Sep-Oct;15(5):46-59. PMID 34548863
- See also: Study Results — https://pubmed.ncbi.nlm.nih.gov/35191173/